CLINICAL TRIAL: NCT00215514
Title: A Pilot Study of Adjuvant Chemoradiation After Resection of Gastric Or Gastroesophageal Junction Adenocarcinoma
Brief Title: Adjuvant Chemoradiation Therapy for Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Charles S. Fuchs, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 00-165
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Stomach Cancer; Gastric Cancer; Gastro-esophageal Junction Cancer
Keywords: adjuvant chemoradiation; GE junction; epirubicin
MeSH Terms: conditions — Stomach Neoplasms | interventions — Epirubicin; Cisplatin; Fluorouracil; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ECF followed by 5-FU/RT followed by ECF (Experimental)
  Interventions: Drug: Epirubicin; Drug: Cisplatin; Drug: 5-Fluorouracil (5-FU); Procedure: Radiation

INTERVENTIONS:
Drug: Epirubicin — Epirubicin (Day 1), Cisplatin (Day 1), 5-FU (Days 1-21)--> One-week rest --> External Beam Radiation Therapy plus 5-FU CI --> Four-week rest --> Epirubicin (Day 1), Cisplatin (Day 1), 5-FU (Days 1-21)--> Epirubicin (Day 1), Cisplatin (Day 1), 5-FU (Days 1-21).
Drug: Cisplatin — Epirubicin (Day 1), Cisplatin (Day 1), 5-FU (Days 1-21)--> One-week rest --> External Beam Radiation Therapy plus 5-FU CI --> Four-week rest --> Epirubicin (Day 1), Cisplatin (Day 1), 5-FU (Days 1-21)--> Epirubicin (Day 1), Cisplatin (Day 1), 5-FU (Days 1-21).
Drug: 5-Fluorouracil (5-FU) — Epirubicin (Day 1), Cisplatin (Day 1), 5-FU (Days 1-21)--> One-week rest --> External Beam Radiation Therapy plus 5-FU CI --> Four-week rest --> Epirubicin (Day 1), Cisplatin (Day 1), 5-FU (Days 1-21)--> Epirubicin (Day 1), Cisplatin (Day 1), 5-FU (Days 1-21).
Procedure: Radiation — Epirubicin (Day 1), Cisplatin (Day 1), 5-FU (Days 1-21)--> One-week rest --> External Beam Radiation Therapy plus 5-FU CI --> Four-week rest --> Epirubicin (Day 1), Cisplatin (Day 1), 5-FU (Days 1-21)--> Epirubicin (Day 1), Cisplatin (Day 1), 5-FU (Days 1-21).

SUMMARY:
The main purpose of this trial is to determine how well patients with gastric or gastroesophageal junction adenocarcinoma respond to chemotherapy with epirubicin, cisplatin and 5-fluorouracil followed by continuous infusion 5-fluorouracil chemotherapy given along with radiation therapy.

DETAILED DESCRIPTION:
* Patients will receive epirubicin and cisplatin intravenously on day 1 of treatment. 5-fluorouracil will be given continuously by intravenous infusion bia a portable ambulatory pump (CADD pump) for 21 days. This cycle of chemotherapy will take 21 days (3 weeks). Once it is complete there will be one week without therapy.
* Once the patient has recovered from any side-effects from the chemotherapy they will start the combination chemoradiation therapy, 5-fluorouracil and radiation. The radiation will be directed to the upper abdomen in the area where the stomach tumor has been located. The radiation therapy will be given five days a week for a total of five weeks. During these five weeks patients will receive 5-fluorouracil continuously by CADD pump.
* After completion of combination chemoradiation therapy there will be a three to four week rest period followed by 2 additional chemotherapy cycles identical to the first chemotherapy cycle.
* The following tests and procedures will be performed: physical examination every 4 weeks except during the chemoradiation therapy when it will be done weekly; blood tests every week during chemotherapy and chemoradiation; CT scans and chest x-rays done before therapy, at the end of therapy, and yearly for 2 years; noninvasive testing to evaluate kidney function before starting the study.
* The program of chemotherapy and radiation therapy will last approximately 30 weeks. After all treatment is completed, patients will return for physical examinations and blood tests every 3 months for 3 years; then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have adenocarcinoma of the stomach or gastroesophageal junction. Adenocarcinomas of the esophagus that are not involving the gastroesophageal junction are not eligible.
* Patients must have had en bloc resection of all known tumor and be at high risk for later failure. The surgical resection must have been done with a curative intent. The stomach, lver, peritoneum, omentum and regional lymph nodes must be evaluated and all identified tumor be resected.
* The surgical specimen, and the pathologic analysis thereof, must be adequate for TNM staging.
* Treatment must begin between day 20 and day 56 after the gastrectomy.
* ECOG performance status of 0,1 or 2
* ANC > 1,500/ul and platelet count >100,000/ul
* Serum creatinine < 1.5mg/dl
* Total bilirubin < 2.0 mg/dl and AST < 3 x ULN
* Estimated caloric intake of 1500K calories per day or greater

Exclusion Criteria:

* Known unresected cancer, microscopic evidence of tumor at the line of resection, noncontiguous resection of tumor, or M1 disease
* Ascites, peritoneal seeding, liver metastasis or extra-abdominal metastasis
* Prior malignancy except for adequately treated basal cell or squamous cell skin cancer, non-invasive carcinoma in situ which has been fully resected, or other cancer for which the patient has been disease free for five years
* Previous chemotherapy or radiotherapy
* Active infectious process
* Pregnant or lactating women
* Myocardial infarction in the past 6 months or prior history of congestive heart failure or significant valvular heart disease
* Uncontrolled serious medical or psychiatric condition
* Grade 2 or greater peripheral neuropathy at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2000-09; Primary Completion 2003-11 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
To assess patient tolerance and toxicity of postoperative adjuvant regimen using epirubicin, cisplatin, and infusional 5-FU before and after a course of radiotherapy among patients with curatively resected gastric or gastroesophageal adenocarcinoma. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles S. Fuchs, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts